CLINICAL TRIAL: NCT01915862
Title: Comparison of Blood Pressure Variability Indices and Ambulatory Arterial Stiffness Index as Prognostic Indicators in the Medium Term Outcome of Acute Ischemic Stroke
Brief Title: Blood Pressure Variability in Acute Ischemic Stroke
Acronym: PREVISE
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: A & D Company Limited (Industry)
Responsible Party: Principal Investigator, Nikolaos Kakaletsis, MD, MSc, Resident in Internal Medicine, AHEPA University Hospital, Aristotle University Of Thessaloniki
Other Study IDs: AUTH-A7399-1862013
Record Dates: First submitted 2013-08-01; First posted 2013-08-05 (Estimated); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Ischemic Stroke
Keywords: Acute ischemic stroke; Blood pressure variability; Ambulatory arterial stiffness index; Ambulatory blood pressure monitoring; Outcome
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is the evaluation and comparison of blood pressure variability indices and ambulatory arterial stiffness index obtained by ambulatory blood pressure monitoring as prognostic indicators in the functional outcome of acute ischemic stroke.

DETAILED DESCRIPTION:
All consecutive patients admitted with acute (within 24 hours after stroke onset) ischemic stroke in three University Hospital of Northern and Central Greece will be included.

Blood pressure measurements are being obtained with ambulatory 24-hour BP monitoring (ABPM) every 20 minutes within 24 hours of admission using automated oscillometric device (TM2430, A&D Company Ltd) during day-time (7:00-22:59) and night-time (23:00-6:59).

Several clinical, laboratory and imaging parameters are prospectively registered. Also, patients' medical history, previous medical treatment and cardiovascular risk factors are registered.

Functional outcome is assessed by the modified Rankin Scale score at 3 months. Also, stroke recurrence and cardiovascular and all-cause mortality will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke
* Admission within 24 after the onset of symptoms

Exclusion Criteria:

* Transient ischemic attack
* Intracerebral hemorrhage
* Subarachnoid hemorrhage
* Cerebral sinus venous thrombosis
* Stroke mimics
* Late admission (>24 hours after stroke onset)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients admitted to Departments of Medicine of three University Hospitals (Thessaloniki, Larissa, Ioannina) with the diagnosis of acute ischemic stroke
Sampling Method: Non-Probability Sample
Enrollment: 353 (Actual)
Dates: Start 2013-08; Primary Completion 2018-05 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale Score (mRS) | Three months (90 days)
  Description (score)
  * No symptoms at all (0)
  * No significant disability despite symptoms; able to carry out all usual duties and activities (1)
  * Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance (2)
  * Moderate disability; requiring some help, but able to walk without assistance (3)
  * Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance (4)
  * Severe disability; bedridden, incontinent and requiring constant nursing care and attention(5)
  * Dead (6)

CONTACTS AND LOCATIONS:
Overall Officials: Apostolos I. Hatzitolios, MD, PhD, Study Director — Aristotle University of Thessaloniki, AHEPA University Hospital
Locations (3):
- Greece (3):
  - Second Department of Internal Medicine, Medical School, University of Ioannina, University Hospital of Ioannina, Ioannina
  - Department of Medicine, Medical School, University of Thessaly, University Hospital of Larissa, Larissa
  - First Propedeutic Department of Internal Medicine, Medical School, Aristotle University of Thessaloniki, AHEPA University Hospital, Thessaloniki

REFERENCES:
- [Background] Kakaletsis N, Ntaios G, Milionis H, Haidich AB, Makaritsis K, Savopoulos C, Berge E, Hatzitolios AI. Prognostic value of 24-h ABPM in acute ischemic stroke for short-, medium-, and long-term outcome: a systematic review and meta-analysis. Int J Stroke. 2015 Oct;10(7):1000-7. doi: 10.1111/ijs.12609. Epub 2015 Aug 18. PMID 26283262
- [Result] Kakaletsis N, Ntaios G, Milionis H, Karagiannaki A, Chouvarda I, Dourliou V, Chytas A, Hatzitolios AI, Savopoulos C. Prognostic significance of 24-h blood pressure and variability indices in the outcome of acute ischaemic stroke. Intern Med J. 2023 Jul;53(7):1137-1146. doi: 10.1111/imj.15834. Epub 2022 Sep 12. PMID 35666577
- [Result] Kakaletsis N, Ntaios G, Milionis H, Protogerou AD, Karagiannaki A, Chouvarda I, Dourliou V, Ladakis I, Kaiafa G, Daios S, Doumas M, Savopoulos C. Time of blood pressure in target range in acute ischemic stroke. J Hypertens. 2023 Feb 1;41(2):303-309. doi: 10.1097/HJH.0000000000003331. Epub 2022 Nov 25. PMID 36583356
- [Result] Kakaletsis N, Ntaios G, Milionis H, Karagiannaki A, Chouvarda I, Dourliou V, Ladakis I, Kaiafa G, Vemmos K, Savopoulos C. Midday Dipping and Circadian Blood Pressure Patterns in Acute Ischemic Stroke. J Clin Med. 2023 Jul 21;12(14):4816. doi: 10.3390/jcm12144816. PMID 37510931
- [Result] Karagiannaki A, Kakaletsis N, Chouvarda I, Dourliou V, Milionis H, Savopoulos C, Ntaios G. Association between antihypertensive treatment, blood pressure variability, and stroke severity and outcomes in acute ischemic stroke. J Clin Neurosci. 2024 Jul;125:51-58. doi: 10.1016/j.jocn.2024.05.014. Epub 2024 May 15. PMID 38754240